CLINICAL TRIAL: NCT00712946
Title: Preoperative Heart Rate Variability and Baroreflex Sensitivity in ASO Patients During Various Sleep Stages
Acronym: Barosleep
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: Turku University Hospital (Other Government); University of Turku (Other); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Dr. Timo Laitio (Timo.Laitio@tyks.fi), Department of Anesthesiology and Intensive Care, Turku University Hospital
Other Study IDs: M1155457
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2010-03

CONDITIONS: Arteriosclerosis Obliterans
MeSH Terms: conditions — Arteriosclerosis Obliterans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Arteriosclerosis obliterans patients undergoing elective vascular surgery
- 2: Healthy age-matched volunteers

SUMMARY:
The goal of this study is to evaluate the possible preoperative predictive value of altered heart rate variability (HRV) and baroreflex sensitivity in different sleep stages for postoperative adverse cardiac events (i.e. arrhythmia or myocardial ischemia needing hospitalization or medication, myocardial ischemia assessed by enzyme release, myocardial infarction, sudden cardiac death, stroke) in arteriosclerosis obliterans patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* ASO
* Elective vascular surgery patient (i.e. infra-inguinal bypass procedure)

Exclusion Criteria:

* Other than sinus rhythm
* Lack of co-operation
* Major surgery less than 3 months preoperatively
* Sleep apnoea
* Dialysis treatment
* CABG less than 3 years earlier

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASO patients admitted to electrive vascualr surgery in Turku University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2006-03; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timo Laitio, MD, PhD, Principal Investigator — Turku University Hospital; Pekka Meriläinen, Prof., Study Director — GE Healthcare, Finland
Locations (1):
- Department of Anesthesiology and Intensive Care, Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Virtanen S, Utriainen KT, Parkkola R, Airaksinen JK, Laitio R, Scheinin H, Hakovirta H, Laitio TT; BAROSLEEP Study Group. White matter damage of the brain is associated with poor outcome in vascular surgery patients with claudication: a pilot study. Eur J Vasc Endovasc Surg. 2014 Dec;48(6):687-93. doi: 10.1016/j.ejvs.2014.08.025. Epub 2014 Oct 1. PMID 25544158
- [Derived] Utriainen KT, Airaksinen JK, Polo O, Laitio R, Pietila MJ, Scheinin H, Vahlberg T, Leino KA, Kentala ES, Jalonen JR, Hakovirta H, Parkkola R, Virtanen S, Laitio TT. Sleep apnoea is associated with major cardiac events in peripheral arterial disease. Eur Respir J. 2014 Jun;43(6):1652-60. doi: 10.1183/09031936.00130913. Epub 2014 Feb 20. PMID 24558173
- [Derived] Utriainen KT, Airaksinen JK, Polo O, Raitakari OT, Pietila MJ, Scheinin H, Helenius HY, Leino KA, Kentala ES, Jalonen JR, Hakovirta H, Salo TM, Laitio TT. Unrecognised obstructive sleep apnoea is common in severe peripheral arterial disease. Eur Respir J. 2013 Mar;41(3):616-20. doi: 10.1183/09031936.00227611. Epub 2012 Jun 14. PMID 22700841